CLINICAL TRIAL: NCT03134209
Title: A Single-center, Phase IV, Randomized, Prospective Study Investigating the Efficacy of Various Wound Closure Devices in Reducing Postoperative Wound Complications
Brief Title: A Study Investigating the Efficacy of Various Wound Closure Devices in Reducing Postoperative Wound Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-02020
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Joint Disease; Arthropathy
Keywords: Monocryl; Dermabond; Polyester mesh; Joint Disease; Arthropathy; Joint Replacement
MeSH Terms: conditions — Joint Diseases | interventions — glycolide E-caprolactone copolymer; octyl 2-cyanoacrylate

STUDY DESIGN:
Intervention Model Description: Zipper surgical skin closure device applied to the most superficial layer of skin following a joint arthroplasty will be compared to two groups: 1) Monocryl + Dermabond 2) Polyester mesh + Dermabond
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Zipper surgical skin closure (Experimental): Zipper surgical skin closure device applied to the most superficial layer of skin following a joint arthroplasty
  Interventions: Device: Zipper surgical skin closure
- Monocryl + Dermabond (Active Comparator): Monocryl suture plus Dermabond is a commonly used combination of wound closure techniques today.
  Interventions: Other: Monocryl + Dermabond
- Polyester mesh + Dermabond (Active Comparator): The polyester plus Dermabond closure techniques combines the OCA topical skin adhesive with a flexible, self-adhesive polyester mesh that has proven to reduce wound cosure times and have a significant greater skin holding strength than skin staples or subcuticular sutures in one study
  Interventions: Other: Polyester mesh + Dermabond

INTERVENTIONS:
Device: Zipper surgical skin closure — The device acts like a scaffold to stabilize the adjacent sides of a wound in order to minimize forces that can disrupt normal healing of the skin.
  Arms: Zipper surgical skin closure
Other: Monocryl + Dermabond — conventional sutures and skin adhesive glue
  Arms: Monocryl + Dermabond
Other: Polyester mesh + Dermabond — conventional sutures and skin adhesive glue
  Arms: Polyester mesh + Dermabond

SUMMARY:
A single-center, phase IV, randomized, prospective study investigating the efficacy of various wound closure devices in reducing postoperative wound complications.

DETAILED DESCRIPTION:
The zipper wound technology is a new wound closure device that is an alternative to the commonly used conventional staples and sutures. The device acts like a scaffold to stabilize the adjacent sides of a wound in order to minimize forces that can disrupt normal healing of the skin. The other treatment groups include monocryl + Dermabond (conventional sutures and skin adhesive glue) and polyester mesh + Dermabond. All products have been FDA approved. A randomized control trial will provide the highest level of evidence without altering the potential risks to the patient as all three wound closure techniques have been found to have comparable complication rates. The three different treatment devices will be administered following the normal standard of care. All three wound closure devices are currently being used at NYULMC. No modifications to the normal standard of practice other than the randomization process will be implemented. Given the nature of the application of the wound closure device, which will be visible to the surgeon at the time of application and the patient postoperatively, the study will not be blinded to either the surgeon or the patient. Prior to discharge, a blinded plastic surgeon will be asked to assess the wound based on comesis and overall quality of wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing joint arthroplasty

Exclusion Criteria:

* Treatment of total joint replacement surgery at an outside institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zipper Surgical Skin Closure | Monocryl + Dermabond | Polyester Mesh + Dermabond
Started | 53 | 54 | 53
Completed | 53 | 54 | 53
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zipper Surgical Skin Closure | Monocryl + Dermabond | Polyester Mesh + Dermabond | Total
Number analyzed (Participants) | 53 | 54 | 53 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.75) | 64.56 (10.37) | 66.51 (8.92) | 65.78 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 36 | 107
  Male | 14 | 22 | 17 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 9 | 24
  Not Hispanic or Latino | 45 | 47 | 44 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 6 | 20
  White | 30 | 30 | 33 | 93
  More than one race | 4 | 0 | 0 | 4
  Unknown or Not Reported | 8 | 12 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 53 | 160

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Pain
Description: The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity along a horizontal line, and this rating is then measured from the left edge. The total range of score is 0-10; the higher the score the worse the pain (0 = no pain, 10 = worst pain imaginable).
Time Frame: 4 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zipper Surgical Skin Closure | Monocryl + Dermabond | Polyester Mesh + Dermabond
Number analyzed (Participants) | 53 | 54 | 53
score on a scale | 4.53 (1.85) | 4.48 (1.78) | 4.54 (1.76)

ADVERSE EVENTS:
Time Frame: 30 days following the last administration of study treatment
Arm/Group | Zipper Surgical Skin Closure | Monocryl + Dermabond | Polyester Mesh + Dermabond
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/54 | 1/53
Other Adverse Events (participants affected / at risk) | 2/53 | 1/54 | 1/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zipper Surgical Skin Closure (N=53) | Monocryl + Dermabond (N=54) | Polyester Mesh + Dermabond (N=53)
Revision Surgery (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zipper Surgical Skin Closure (N=53) | Monocryl + Dermabond (N=54) | Polyester Mesh + Dermabond (N=53)
Wound Drainage (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03134209/Prot_SAP_000.pdf